CLINICAL TRIAL: NCT00229788
Title: Impact of Race and Re-Transplantation in Childhood: Analysis of Data From the United Network of Organ Sharing
Brief Title: Impact of Race and Re-Transplantation
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05.018
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Orthotopic Heart Transplantation
Keywords: orthotopic heart transplantation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
For children who develop graft failure following cardiac transplantation, retransplantation is often considered. While some centers have reported equivalent results for retransplantation as compared to primary transplantation, this strategy remains controversial. We seek to examine outcomes following re-transplantation in children and identify risk factors for mortality. In addition, adult African-Americans have been reported to have lower survival following heart and other solid-organ transplantation. The relationship of recipient race to survival following pediatric heart transplantation has not previously been reported.

DETAILED DESCRIPTION:
Objective 1: For children who develop graft failure following cardiac transplantation, retransplantation is often considered. While some centers have reported equivalent results for retransplantation as compared to primary transplantation, this strategy remains controversial. We seek to examine outcomes following re-transplantation in children and identify risk factors for mortality.

Objective 2: Adult African-Americans have been reported to have lower survival following heart and other solid-organ transplantation. The relationship of recipient race to survival following pediatric heart transplantation has not previously been reported.

Methods: We would like to review the United Network for Organ Sharing database. We plan on reviewing database records of heart transplantation subjects <18 years of age from 1987 to 2004. Indications for retransplantation and patient race characteristics will be collected and evaluated. Analysis will be performed using proportional hazards regression controlling for other potential risk factors. The contribution economic disparity, insurance status and HLA mismatching to disparities in outcome will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* orthotopic heart transplantation
* < 18 years of age

Exclusion Criteria:

-

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States